CLINICAL TRIAL: NCT04427943
Title: Outcome After Revisions of Infected Knee Arthroplasties - a Prospective Multicenter Cohort Study
Brief Title: Outcome After Revisions of Infected Knee Arthroplasties
Acronym: RIKA
Status: Active, not recruiting | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Martin Lindberg-Larsen, Principal investigator, Odense University Hospital
Other Study IDs: S-20170108/69984
Record Dates: First submitted 2020-01-08; First posted 2020-06-11 (Actual); Last update posted 2024-12-11 (Actual); Status verified 2024-12

CONDITIONS: Periprosthetic Knee Infection
Keywords: infection; knee arthroplasty; surgical treatment; patient reported outcome
MeSH Terms: conditions — Infections | interventions — Reoperation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (1):
- RIKA cohort: patients with periprosthetic knee joint infection scheduled for revision knee arthroplasty surgery
  Interventions: Procedure: revision surgery

INTERVENTIONS:
Procedure: revision surgery — The intervention is the planned revision surgery according to local guidelines.

SUMMARY:
A prospective multicenter cohort study on all types of revision knee arthroplasty procedures performed due to infection.

DETAILED DESCRIPTION:
A prospective multicenter cohort study on all types of revision knee arthroplasty procedures performed due to infection.

Most previous studies investigating outcomes after revisions of infected knee artrplasties are single-center studies and retrospective. The study group has previously investigated outcome of the surgical treatment of infected knee arthroplasties in Denmark based on nationwide data from Danish registries. These studies revealed that the risk of treatment failure causing re-revision or mortality was 30-40% in Denmark.

Based on these findings, an ongoing randomized controlled trial "one-stage versus two-stage revisions of the infected knee arthroplasty" (ClinicalTrials.gov ID: NCT03435679) has been initiated by the study group in Febuary 2018. It has been possible to include 20% of the patients with surgically demanding periprosthetic knee infections from the including centres in this randomized trial due to in- and exclusions criteria. Hence, the investigators wish to include the remaining patients with periprosthetic knee joint infection in a prospective cohort study in order to obtain high quality prospective data on function, quality of life and complications after all types of surgical procedures performed due to periprosthetic knee joint infection. Based on these data it will be possible to evaluate the surgical treatment overall and it will be possible to evaluate whether the patients included in the randomized trial are representative.

Study aim:

To present patient reported outcome and postoperative complications after all types of surgical procedures performed due to periprosthetic knee infection. Furthermore, to analyze the role of potential risk factors (patient comorbidity, microbiological diagnosis, surgical intervention, antibiotic treatment, duration of symptoms) on outcome of the patients.

ELIGIBILITY:
Inclusion Criteria:

* Clinical signs of periprosthetic knee joint infection and indication for revision surgery
* Speak and understand Danish and have given informed consent

Exclusion Criteria:

* Participation in "one-stage versus two-stage revisions of the infected knee arthroplasty"

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with periprosthetic knee joint infection requiring revision surgery.
Sampling Method: Non-Probability Sample
Enrollment: 350 (Estimated)
Dates: Start 2020-01-01 (Actual); Primary Completion 2025-11 (Estimated); Study Completion 2026-11 (Estimated)

PRIMARY OUTCOMES:
Change in Oxford Knee Score (Area Under Curve (AUC) from preoperatively to 12 months postoperatively) | Measured preoperatively 6 weeks, 3, 6, 9, 12 months postoperatively
  Change in Oxford Knee Score from preoperatively to 12 months postoperatively measured as Area Under Curve. Oxford Knee Score ranges from 0 to 48, 48 = best score.

SECONDARY OUTCOMES:
Change in Oxford Knee Score (Area Under Curve, AUC from preop. to 12 months postop.) | Time Frame: Measured preoperatively, 6 weeks, 3, 6, 9, 12, 18 and 24 months postoperatively
  Change in Oxford Knee Score from preoperatively to 24 months postoperatively measured as Area Under Curve. Oxford Knee Score ranges from 0 to 48, 48 = best score.
Change in EuroQol five-dimensional descriptive system (EQ-5D-5L) from preop to 24 months postop. | Measured preoperatively, 6 weeks, 3, 6, 9, 12, 18 and 24 months postoperatively.
  Quality of life questionnaire
Number of participants re-revised (re-revision rate) | 2 year postoperatively
  Number of patients re-revised due to infection and other causes within 2 years postoperatively.
Number of participants dying (mortality rate) | 2 years postoperatively
  Number of participants dying within 2 years posoperatively
Number of participants readmitted (readmission rate) | 90 days postoperatively
  Number of participant readmitted within 90 days postoperatively

CONTACTS AND LOCATIONS:
Overall Officials: Martin Lindberg-Larsen, MD, PhD, Principal Investigator — Odense University Hospital
Locations (8):
- Denmark (8):
  - Aalborg University Hospital, Aalborg
  - Bispebjerg Hospital, Copenhagen
  - Hvidovre, Copenhagen
  - Rigshospitalet, Copenhagen
  - Horsens Hospital, Horsens
  - Næstved Hospital, Næstved
  - Odense Universitets Hospital, Odense
  - Vejle Hospital, Vejle

IPD SHARING:
Plan to Share IPD: No
According to local interpretation of GDPR. Blided data can be provided upon request.

REFERENCES:
- [Background] Lindberg-Larsen M, Pitter FT, Voldstedlund M, Schroder HM, Bagger J. Microbiological diagnosis in revision of infected knee arthroplasties in Denmark. Infect Dis (Lond). 2017 Nov-Dec;49(11-12):824-830. doi: 10.1080/23744235.2017.1350878. Epub 2017 Jul 8. PMID 28691647
- [Background] Lindberg-Larsen M, Jorgensen CC, Bagger J, Schroder HM, Kehlet H. Revision of infected knee arthroplasties in Denmark. Acta Orthop. 2016 Aug;87(4):333-8. doi: 10.3109/17453674.2016.1148453. Epub 2016 Feb 22. PMID 26900908
- [Derived] Lindberg-Larsen M, Odgaard A, Fredborg C, Schroder HM; One-stage vs Two-stage Collaboration Group. One-stage versus two-stage revision of the infected knee arthroplasty - a randomized multicenter clinical trial study protocol. BMC Musculoskelet Disord. 2021 Feb 12;22(1):175. doi: 10.1186/s12891-021-04044-8. PMID 33579256